CLINICAL TRIAL: NCT01849250
Title: A Multicenter Phase II Study of Docosahexaenoic Acid (DHA) in Patients With a History of Breast Cancer, Premalignant Lesions, or Benign Breast Disease
Brief Title: Study of Docosahexaenoic Acid (DHA) in Triple Negative Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2013-00859; NCI-2013-00859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-474; 12-267; N01-CN-2012-00034; DFCI:12- 474 (Other: Dana-Farber Cancer Institute (DFCI)); AAAK6752; MSKCC-12-267 (Other: Memorial Sloan Kettering Cancer Center (MSK or MSKCC)); H-33017; CUMC: AAAK6752; 2011-0766 (Other: MD Anderson Cancer Center (MDA or MDACC)); MDA10-16-01 (Other: DCP); N01CN00034 (NIH); N01CN35159 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Benign Breast Neoplasm; Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Lobular Breast Carcinoma In Situ; Paget Disease of the Breast; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Paget's Disease, Mammary; Breast Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Docosahexaenoic Acid) (Experimental): Docosahexaenoic Acid orally twice a day (PO BID) for 12 weeks.
  Interventions: Drug: Docosahexaenoic Acid
- Arm II (placebo) (Placebo Comparator): Placebo orally twice a day (PO BID) for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Docosahexaenoic Acid — Given PO
  Other Names: Fatty Acid 22:6
  Arms: Arm I (Docosahexaenoic Acid)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies how well docosahexaenoic acid works in preventing recurrence in breast cancer survivors. Docosahexaenoic acid supplement may prevent recurrence in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether treatment with docosahexaenoic acid (DHA) for 12 weeks at 1000 mg twice daily as compared to placebo reduces normal breast tissue levels of tumor necrosis factor-alpha (TNF-alpha) in overweight and obese patients with a history of stage I-III invasive breast cancer, ductal carcinoma in situ (DCIS), Paget's disease, lobular carcinoma in situ (LCIS), or proliferative benign breast disease.

SECONDARY OBJECTIVES:

I. To investigate the effect of DHA at 1000 mg twice daily on tissue biomarkers

* Change from the baseline in cyclooxygenase-2 (COX-2)/interleukin-1-beta (IL-1beta)/aromatase measured by quantitative real-time polymerase chain reaction (PCR).
* Change from the baseline in crown-like structures of the breast (CLS-B) measured by immunohistochemical techniques for cluster of differentiation (CD)68.
* Change from baseline in CLS-B index determined as follows: ([number of slides with evidence of at least one CLS-B]/[total number of slides examined]).
* Change from baseline in CLS-B/cm^2 defined as the number of CLS-B/cm^2. II. Evaluate age as a predictor of CLS-B and inflammatory biomarkers (TNF-alpha/COX-2/IL-1beta) at baseline and over the time of treatment.

III. Evaluate red blood cell (RBC) fatty acid level as a surrogate of compliance.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive docosahexaenoic acid orally (PO) twice daily (BID) for 12 weeks.

ARM II: Patients receive placebo PO BID for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a history of histologically-confirmed stage I-III invasive breast cancer or ductal carcinoma in situ (DCIS), Paget's disease, lobular carcinoma in situ (LCIS), or proliferative benign breast disease
* No evidence of disease (in situ or invasive cancer that would normally be treated by resection) at trial entry as determined by the investigator
* >= 6 months from all previous breast cancer treatment (including surgery for invasive cancer, chest wall radiotherapy, chemotherapy, trastuzumab and endocrine therapy)
* Participants must have a body mass index (BMI) >= 25, defined as (weight in kilograms/[height in meters]^2)
* Participants must have adequate accessible breast tissue as determined by the treating physician, consisting of one breast unaffected by invasive cancer, which has not been radiated; a history of prior pre-invasive breast cancer or benign biopsy of this breast will be permitted
* Daily DHA consumption =< 200 mg/day in the month prior to screening estimated by an abbreviated DHA food frequency questionnaire
* Mammogram within no more than 6 months prior to the date of informed consent (normal/benign Breast Imaging-Reporting and Data System [BI-RADS] 1 or 2) and no further routine breast imaging planned during the course of the study (12 weeks DHA/placebo)
* Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 75,000/uL
* White blood cells >= 3,000/uL
* Hemoglobin >= 10 g/dL
* Total bilirubin within 1.5 times the institution's upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) within 1.5 times the institution's ULN
* Serum creatinine within 1.5 times the institution's ULN
* Pregnant women will be excluded; for women of childbearing potential; negative pregnancy testing within 72 hours prior to or on study visit #1 (day 0) and willingness to use adequate contraception during the study intervention OR post-menopausal defined as any one of the following 1) prior hysterectomy, 2) absence of menstrual period for 1 year in the absence of prior chemotherapy or 3) absence of menstrual period for 2 years in women with a prior history of chemotherapy exposure who were pre-menopausal prior to chemotherapy
* Willingness to comply with all study interventions and follow-up procedures including the ability to swallow the study drug
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any type of active invasive cancer (excluding breast and non-melanoma skin cancer) within the preceding 18 months
* A history of histologically-confirmed bilateral invasive breast cancer
* Bilateral mastectomy
* Prior history or evidence of metastatic breast cancer
* Prior radiation therapy to the contralateral (unaffected) breast
* Prior history of contralateral (unaffected) breast augmentation with breast implant placement
* History of daily use of aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) in the week preceding study entry
* History of DHA supplementation > 200 mg/day in the month preceding study entry
* History of autoimmune disorder or any illness that requires therapy with chronic steroids or immunomodulators
* History of therapeutic doses of anticoagulants including warfarin and low molecular weight heparin (e.g. for prior deep venous thrombosis and pulmonary embolism) in the preceding year
* Participants may not be receiving any other investigational agents during the study
* Women who have received cancer surgery, chemotherapy, biological therapy (e.g., trastuzumab), or radiotherapy for the treatment of any cancer within 6 months of study participation
* Women who are receiving endocrine therapy for breast cancer treatment or chemoprevention including tamoxifen, letrozole, anastrozole, fulvestrant, or exemestane at the time of screening
* Individuals with severe underlying chronic illness, such as uncontrolled diabetes; ongoing or active infection, psychiatric illness or social situations which in the opinion of the investigator would interfere with study participation
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DHA or corn/soy oil in placebo agent
* Pregnant, breastfeeding, or women of childbearing potential unwilling to use a reliable contraceptive method

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Gucalp, Principal Investigator — Memorial Sloan Kettering Cancer Center; Powel H. Brown, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 1 ,2013 to December 31, 2015. All recruitment done in medical settings.
Pre-assignment Details: Of 65 participants enrolled, one was not eligible thus excluded from the study.
Groups:
- Placebo: Placebo orally twice a day for 12 weeks.
- Docosahexaenoic Acid (DHA): Docosahexaenoic Acid 1000 mg orally twice a day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 32 | 32
Completed | 25 | 29
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not Evaluable | 5 | 3
Not completed — Screen Failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Docosahexaenoic Acid: DHA 1000 mg orally twice a day for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Docosahexaenoic Acid | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [52 to 62] | 59.5 [51 to 63] | 59 [52 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 22 | 25 | 47
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 27 | 28 | 55
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Normal Breast Tissue Expression of Tumor Necrosis Factor Alpha (TNF-alpha) Levels
Description: Differences in normal breast tissue levels of TNF-α 12 weeks post-treatment relative to pre-treatment for active treatment and placebo arm, compared using analysis of covariance where the post-treatment measurements were used as a dependent variable and the pretreatment measurements were included as a covariate in the analysis. For the primary study end-point TNF-α levels will be measured by quantitative real-time PCR (mRNA essays) on extracted RNA from breast core biopsies. Relative expression determined using the Computed Tomography (ΔΔCT) analysis protocol.
Time Frame: Baseline to 12 weeks
Population: 6 participants in the Placebo group and 1 participant in the DHA group were not evaluable due to tissue was not available quantitative RT-PCR.
Measure: Mean (Standard Deviation); unit: Log Transformed Relative ExpressionLevel
Groups:
- Docosahexaenoic Acid: Docosahexaenoic Acid (DHA) 1000 mg orally twice a day for 12 weeks.
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 26 | 31
Log Transformed Relative ExpressionLevel
  Baseline | 0.26 (0.93) | 0.08 (0.78)
  Post-Treatment | 0.06 (0.92) | 0.16 (0.95)
  Post-treatment vs. Baseline Change | -0.22 (1.19) | 0.08 (0.99)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .50, ANCOVA

2. Secondary Outcome: Number of Participants With Crown-like Structures of the Breast (CLS-B) at Baseline and Post-treatment
Description: An indicator of whether a subject is detected with CLS-B or not.
Time Frame: Baseline to 12 weeks
Population: 4 participants on the placebo arm and 1 participant on the DHA arm did not have a post treatment biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 28 | 31
Participants
  Baseline | 2 | 4
  Post-treatment | 3 | 3
  Positive both Baseline and Post-treatment | 2 | 0

3. Secondary Outcome: Absolute Change in CLS-B/cm^2 Adjusted for the Pre-treatment Measurements
Description: To assess the severity of CLS-B using the following formula: number of CLS-B/cm^2. The absolute change in the CLS-B/cm^2 calculated according to the formula; Change in CLS-B/cm^2 = (post-treatment CLS-B/cm^2) - (pre-treatment CLS-B/cm^2).
Time Frame: Baseline to 12 weeks
Population: Data were not collected.
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Breast Tissue Cox 2 mRNA Levels at Baseline and 12 Weeks
Description: Biomarkers COX-2 are measured by quantitative real-time PCR. Differences between active treatment and placebo arm for each biomarker will be compared using analysis of covariance where the post treatment measurements will be used as a dependent variable and the pretreatment measurements will be included as a covariate in the analysis.
Time Frame: Baseline to 12 weeks
Population: Participants with adequate RNA available were analyzed.
Measure: Mean (Standard Deviation); unit: relative expression level
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 14 | 23
relative expression level
  Baseline COX-2 | 0.49 (1.35) | 0.31 (0.97)
  Post-Treatment COX-2 | -0.11 (1.30) | 0.22 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Docosahexaenoic Acid; Test type: Superiority; p = .19, ANCOVA

5. Secondary Outcome: Mean Difference in the Breast Tissue IL- Beta mRNA Levels of Tissue Biomarkers
Description: Biomarkers IL-1Beta are measured by quantitative real-time PCR. Differences between active treatment and placebo arm for each biomarker will be compared using analysis of covariance where the post treatment measurements will be used as a dependent variable and the pretreatment measurements will be included as a covariate in the analysis.
Time Frame: Baseline to 12 weeks
Population: Participants with adequate RNA available were analyzed.
Measure: Mean (Standard Deviation); unit: relative expression level
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 26 | 31
relative expression level
  Baseline IL-Beta | 0.62 (2.00) | 0.28 (1.50)
  Post-treatment IL-Beta | 0.23 (2.06) | 0.19 (2.07)
Statistical Analysis 1: Comparison: Placebo vs Docosahexaenoic Acid; Test type: Superiority; p = .52, ANOVA

6. Secondary Outcome: Mean Difference in the Breast Tissue Aromatase mRNA Levels of Tissue Biomarkers
Description: Biomarkers Aromatase are measured by quantitative real-time PCR. Differences between active treatment and placebo arm for each biomarker will be compared using analysis of covariance where the post treatment measurements will be used as a dependent variable and the pretreatment measurements will be included as a covariate in the analysis.
Time Frame: Baseline and 12 weeks
Population: Participants with adequate RNA available were analyzed.
Measure: Mean (Standard Deviation); unit: relative expression level
Arm/Group | Placebo | Docosahexaenoic Acid
Number analyzed (Participants) | 22 | 30
relative expression level
  Baseline Aromatase | -0.38 (1.93) | 0.13 (2.38)
  Post-treatment Aromatase | -0.59 (2.13) | 0.06 (1.89)
Statistical Analysis 1: Comparison: Placebo vs Docosahexaenoic Acid; Test type: Superiority; p = .12, ANCOVA

7. Secondary Outcome: Red Blood Cell (RBC) Fatty Acid Level as a Surrogate of Compliance
Description: Whole blood samples collected for red blood cell fatty acid analyses at baseline and week 12 (+ 2 weeks). RBC fatty acid composition analyzed by gas chromatography (GC) with flame ionization detection.
Time Frame: Baseline and week 12
Population: Available blood samples.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 28 | 30
percentage
  Baseline Omega3 index | 5.03 (1.65) | 5.01 (1.13)
  Baseline DHA level | 4.53 (1.5) | 4.47 (0.98)
  Post-Treatment Omega3 index | 4.92 (1.68) | 11.95 (1.35)
  Post-Treatment DHA level | 4.41 (1.48) | 11.2 (1.33)
  Post Treatment v. Baseline Change Omega3 index | -0.10 (.068) | 6.99 (1.43)
  Post Treatment v. Baseline Change DHA level | -0.12 (0.59) | 6.78 (1.42)

ADVERSE EVENTS:
Time Frame: Adverse events collected over 12 weeks of treatment.
Groups:
- Docosahexaenoic Acid: Docosahexaenoic Acid 1000 mg orally twice a day for 12 weeks.
Arm/Group | Placebo | Docosahexaenoic Acid
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 17/32 | 15/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Docosahexaenoic Acid (N=32)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (2)
Dyspepsia - Heart Burn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other: Burping (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrointestinal disorders - Other: Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other: Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Heart failure, Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - other, Poison Ivy Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less